CLINICAL TRIAL: NCT01704742
Title: A Prospective Clinicopathological Cohort Study of Lymphoproliferative Diseases at Kenyatta National Hospital in Nairobi, Kenya
Brief Title: Prospective Study of Lymphoproliferative Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Protocol not considered a clinical trial for registration purposes; no subjects enrolled to date pending further grant funding
Sponsor: West Virginia University (Other)
Collaborators: Kenyatta National Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: WVU1411
Record Dates: First submitted 2012-10-03; First posted 2012-10-11 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Kenya; Epstein Barr Virus (EBV); Human Immunodeficiency Virus (HIV); Kaposi's Sarcoma Herpes Virus (KSHV)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Epstein-Barr Virus Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, blood plasma and serum upon consent and suitability of sample preparation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
This study will help researchers learn more about non-Hodgkin's lymphoma and Hodgkin's lymphoma and how it is treated in Kenya. Researchers want to see if having certain viruses like Epstein Barr Virus (EBV), Human Immunodeficiency Virus (HIV), and Kaposi's Sarcoma Herpes Virus (KSHV) affects lymphoma. Patients in Kenya who agree to be in this study will let the resesarchers look at their medical record, follow their normal cancer care, and have blood drawn to look at different proteins and viruses. Researchers would also like to look at part of the original tumor that was taken out of each patient. Some of these samples will be stored at Kenyatta National Hospital and research will be done on them later. This study does not involve any change in treatment, but only allows the study team to follow how a patient in Kenya with lymphoma is treated.

DETAILED DESCRIPTION:
Comprehensive prospective cohort study of lymphoproliferative diseases in Nairobi, Kenya.

ELIGIBILITY:
Inclusion Criteria:

* All subjects regardless of age, sex or HIV serostatus must have biopsy-proven non-Hodgkin's (NHL), including primary effusion lymphoma, Hodgkin's lymphoma (HD) or other lymphoproliferative disorder (e.g., Castleman's disease) with measurable or evaluable stage I through IV disease.

[Note: Lymphomas will be categorized on the basis of current WHO classification scheme, but it is recognized that initial pathological categorization at time of study enrollment will more than likely be classified or graded as low-, intermediate-, or high-grade lymphoma by Working Formulation criteria. This is the current standard of practice in Kenya.]

* All subjects must receive some form of systemic chemotherapy. Subjects not receiving chemotherapy of any kind are not eligible. Subjects must not have had any prior chemotherapy for lymphoma.
* Subjects may have received prior radiotherapy for localized stage I or stage II disease that is clearly documented to have progressed beyond initial radiotherapy ports.
* All subjects must give written informed consent to participate on study. In Kenya, a child is considered < 18 years of age and an adult ≥ 18 years of age. All children will have their parental or legal guardian provide consent.. Children between the ages of 7 and < 18 years old should be given the opportunity to provide their assent. For children between the ages of 7 and 11 years old this should be done using the parental consent form assent statement. For children > 11 years old assent should be documented using the IRB approved assent form.

Exclusion Criteria:

* Subjects who do not fulfill the criteria as listed in Sections 3.1.1 through 3.1.4 are ineligible.
* Subjects who received prior chemotherapy (i.e., first-line treatment) or are not receiving any chemotherapy for their non-Hodgkin's (NHL) or Hodgkin's lymphoma (HD) are ineligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at Kenyatta National Hospital in Kenya being treated for non-Hodgkin's lymphoma or Hodgkin's lymphoma.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine the spectrum and natural history of lymphoproliferative disorders in Nairobi, Kenya | 2.5 Years
  To determine the spectrum and natural history of lymophoproliferative disorders in Nairobi, Kenya by prospectively recruiting subjects with biopsy-proven malignant lymphoma including non-Hodgkin's and Hodgkin's lymphoma regardless of age, sex and HIV-serostatus (cohort study), who are seen at the Kenyatta National Hospital for treatment.

SECONDARY OUTCOMES:
To perform a comprehensive clinicopathological study in these subjects. | 2.5 Years
  To perform a comprehensive clinicopathological study in these subjects with complete virological, immunophenotypic, and molecular characterization of retrieved tumor tissues and peripheral blood samples for purposes of identifying prognostic and predictive biomarkers of clinical outcome (i.e. treatment response, freedom from disease progression, and overall survival) in which to begin to frame pragmatic, risk-adapted therapeutic interventions suitable for the resource constrained setting in sub-Saharan Africa.
Companion R01 proposal: Clinicopathological Cohort Study of EBV-Associated Lymphomas in Kenya | To be submitted next 6 months to 1 year
  * Aim 1: Determine the tissue biomarkers of EBV infection in AIDS-related lymphomas (ARL) in Kenya
  * Aim 2: Compare the pattern of EBV persistence in patients with EBV+ and EBV- lymphoma
  * Aim 3: Determine predictors of treatment outcome in AIDS-related lymphomas (ARL)

CONTACTS AND LOCATIONS:
Overall Officials: Scot C Remick, MD, Principal Investigator — West Virginia University; Walter O Mwanda, MD, Principal Investigator — Kenyatta National Hospital
Locations (2):
- West Virginia University Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States
- Kenyatta National Hospital (University of Nairobi), Nairobi, Kenya

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] World Health Organization. Cancer. Fact Sheet No. 297, February 2011. Available at http://www.who.int/mediacentre/factsheets /fs297/en/index.html. Accessioned March 28, 2011.
- [Background] World Health Organization. The Global Burden of Disease: 2004 Update. Geneva: WHO, 2008.
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, and Parkin DM. Globocan 2008: cancer incidence and mortality worldwide. Lyon: International Agency for Research on Cancer, 2010. Available at: http://www.iarc/fr/. Accessioned March 28, 2011.
- [Background] Remick SC. Responding to the global cancer burden through partnerships. In: Am. Soc. Clin. Oncol. Ed. Book 2009; 670-4.